CLINICAL TRIAL: NCT06044376
Title: The Consumption Effect of Formula Milk With Triple Bifidobacteria Strains (Bifidobacterium Longum BB536, Bifidobacterium Breve M-16V, and Bifidobacterium Longum Subsp. Infantis M-63) on Fecal Quality and Metabolites in Healthy Children
Brief Title: Ingestion Effect of Formula Milk With Triple Bifidobacteria Strains on Fecal Quality and Metabolites in Healthy Children
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gadjah Mada University (Other)
Collaborators: PT Kalbe Farma Tbk (Industry); Morinaga Milk Industry Co., LTD (Industry)
Responsible Party: Principal Investigator, Endang Sutriswati Rahayu, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PUIPTProbiotikUGM_P002
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Children, Only
Keywords: Children; Fecal sample; Triple Bifidobacterium strains; Probiotic; Formula milk; Indonesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Active Comparator): During the baseline period, all participants consumed milk formula without any addition of probiotics three servings per day for 14 days. One serving of milk formula consists of 36 gram that is diluted in 180 mL lukewarm water.
  The participants in the probiotic group consumed milk formula added with triple Bifidobacterium strain containing Bifidobacterium longum BB536 (6.9 x 10^7 CFU/serving), Bifidobacterium breve M16-V (6.9 x 10^7 CFU/serving), Bifidobacterium longum subsp. infantis M-63 (6.9 x 10^7 CFU/serving). The milk formula is consumed three servings per day for 90 days during the intervention period. One serving of milk formula consists of 36 gram that is diluted in 180 mL lukewarm water.
  Interventions: Combination Product: Formula milk with triple Bifidobacterium probiotic strain
- Placebo Group (Placebo Comparator): During the research period (both baseline and intervention period), all participants consumed milk formula without any addition of probiotics three servings per day for 104 days. One serving of milk formula consists of 36 gram that is diluted in 180 mL lukewarm water.
  Interventions: Other: Formula milk

INTERVENTIONS:
Combination Product: Formula milk with triple Bifidobacterium probiotic strain — Formula milk with triple Bifidobacterium strain containing Bifidobacterium longum BB536 (6.9 x 10^7 CFU/serving), Bifidobacterium breve M16-V (6.9 x 10^7 CFU/serving), Bifidobacterium longum subsp. infantis M-63 (6.9 x 10^7 CFU/serving).
  Arms: Probiotic Group
Other: Formula milk — Formula milk without any addition of probiotic strain
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to compare healthy children between 1 to 3 years old. The main question it aims to answer is

1. Is there an effect towards fecal quality after consuming milk formula supplemented with the triple Bifidobacteria strains (Bifidobacterium longum BB536, Bifidobacterium breve M-16V, and Bifidobacterium longum subsp. infantis M-63)?
2. Is there an effect towards short-chain fatty acid composition after consuming milk formula supplemented with the triple Bifidobacteria strains (Bifidobacterium longum BB536, Bifidobacterium breve M-16V, and Bifidobacterium longum subsp. infantis M-63)?
3. Is there an effect towards clinical profile after consuming milk formula supplemented with the triple Bifidobacteria strains (Bifidobacterium longum BB536, Bifidobacterium breve M-16V, and Bifidobacterium longum subsp. infantis M-63)?

The clinical trial period started off with all the participants consuming a milk formula three times a day, for 14 days as a baseline period. Afterwards, the participants were randomly assigned to one of two groups: probiotic and placebo. Following the baseline period, participants in the probiotic group consumed formulated milk supplemented with the triple Bifidobacteria strains, while the placebo group ingested the same formulated milk without adding triple Bifidobacteria strains for 90 days.

Researchers will compare the probiotic and placebo groups to see if there are any effects towards the fecal quality, short-chain fatty acid level and clinical profile after consuming the milk formula.

DETAILED DESCRIPTION:
This clinical trial is a study of 3 strains of Bifidobacterium was conducted in infants aged 1-3 years in Indonesia. The general objective of this study was to determine the benefits of combined supplementation of Bifidobacteria strains (B. longum BB536, B. breve M-16V, and B. longum subsp. infantis M-63) in healthy children aged 1-3 years. The study is conducted for 104 days with a baseline period of 14 days and continued with an intervention period of 90 days. Participants is divided into two groups, which are the intervention group and the placebo group. The study will be conducted using a double-blind randomized, placebo-controlled trial design. A total of 100 participants will be selected based on inclusion and exclusion criteria.

During the screening period (day 0), socialization of the research and signing of informed consent will be carried out for participants who are willing to participate. Participants were asked not to consume fermented milk products, probiotics and prebiotic fortified food/drinks while participating in research activities.

During the baseline period (Day 14), the participants were asked to consume control milk and, represented by their parents, were also asked to fill out research diaries in the form of diet records, records of probiotic products and prebiotic fortified food/drinks consumed, type and frequency of bowel movements, health complaints felt (discomfort, headaches, stomachaches, respiratory tract-related illnesses and fever), medication consumption records, days where the participants refused to eat. Participants were asked to collect research documents and collect stool samples on day 14 +/- 1.

During the intervention period, from day 15 to day 104, participants consumed 36 grams of the test product or placebo dissolved in 180 ml per serving with a consumption frequency of 3 times per day. Product consumption will be recorded in the product consumption logbook and on the subject's diary record form. Once every 2 weeks a health profile measurement (weight, height, arm circumference, head circumference, skinfold thickness) and sleep quality will be measured. Participants were asked to collect research documents and stool samples on day 104 +/- 1 with the same procedure as in the baseline period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 - 36 months
* Normal nutritional status (z-score height-for-age or z-score weight-for-height: -2 SD < X < 2 SD)
* Has no dairy allergies
* Does not consume breastmilk anymore during the intervention period
* Willing to participate through the whole research period
* Obtain consent from parents or guardians by signing the informed consent form

Exclusion Criteria:

* Has a history of lactose intolerance, congenital and chronic diseases including irritable bowel syndrome, etc.
* Receive antibiotic or other probiotic supplementation during the 14 day of baseline period.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-11-09 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Fecal characteristics | Before and after intervention period (day 13 and day 105)
  Observed the shape, color and consistency of fecal samples that will be combined to be reported as fecal type according to the Bristol Stool Chart
Fecal pH | Before and after intervention period (day 13 and day 105)
  The pH of obtained fecal samples were measured using potential of hydrogen (pH) meter
Bacterial colony characteristics | Before and after intervention period (day 13 and day 105)
  From the fecal samples obtained, direct plating using the selective media for Bifidobacterium (Bifidobacterium Selective Medium or BSM) and Enterobacteriaceae (MacConkey Agar) is conducted. Colony bacterial characterization is based on the cell morphology and Gram strain characteristics under the microscope.
Bifidobacterium's cell count | Before and after intervention period (day 13 and day 105)
  The cell number is a total of Bifidobacteria cells obtained from DNA extraction of stool samples counted using quantitative PCR (qPCR). Cell count will be expressed in colony forming unit per gram (CFU/g).
Enterobactericaeae's cell count | Before and after intervention period (day 13 and day 105)
  The cell number is a total of Enterobacteriaceae's cells obtained from DNA extraction of stool samples counted using quantitative PCR (qPCR). Cell count will be expressed in colony forming unit per gram (CFU/g)
Short chain fatty acids analysis | Before and after intervention period (day 13 and day 105)
  The analysis includes the measurement of acetate, propionate, and butyrate. The analysis uses gas chromatography method.
Biomarker of immune systems | Before and after intervention period (day 13 and day 105)
  The analysis on immune systems' biomarker uses the fecal water obtained from diluting the fecal samples into phosphate buffer. The fecal water is then added with protease inhibitor to keep fecal samples stable during the analysis. The immune system analyzed are interleukin 6 (IL6), interleukin 8 (IL8), interleukin 10 (IL10) and secretory immunoglobulin A (SIgA). All immune systems are read using the enzyme-linked Immunosorbent Assay (ELISA) Reader BioRad iMark.

SECONDARY OUTCOMES:
Defecation frequency records | Everyday during the research period (104 days)
  Participants, represented by their parents or guardian, record their defecation frequency in a daily record.
Dietary pattern records | Four days every two weeks, consists of two weekdays and two weekend days during the research period
  Participants, represented by their parents or guardian, record their dietary patterns in a daily record. The dietary pattern recorded includes type and portion of the foods, snacks and beverages.
Health complaint and medical records | Everyday during the research period (104 days)
  Participants, represented by their parents or guardian, record their health complaint and medical records in a daily record.
Health profile record | Before and after intervention period (day 13 and day 105)
  Participants, represented by their parents or guardian, filled a questionnaire about recent respiratory health conditions.
Gastrointestinal disorder record | Before and after intervention period (day 13 and day 105)
  Participants, represented by their parents or guardian, filled a questionnaire about recent gastrointestinal health conditions.
Sleep quality | Before and after intervention period (day 13 and day 105)
  Participants, represented by their parents or guardian, filled a questionnaire about recent history of the participant's sleep quality.
Behaviour assesment | Before and after intervention period (day 13 and day 105)
  Participants, represented by their parents or guardian, filled a questionnaire about how the participants behave especially how they express their emotions.
Development screening | Before and after intervention period (day 13 and day 105)
  Participants, represented by their parents or guardian, filled a questionnaire about recent gastrointestinal health conditions. The Ages and Questionnaires (ASQ-3) were used based on the participant's current age.
Psychosocial problems | Before and after intervention period (day 13 and day 105)
  Participants, represented by their parents or guardian, filled a questionnaire about possible psychosocial problems. The Pediatric Symptom Checklist (PSC) was used for this measure.
Weight | Once every two weeks for 105 days
  The participants were measured for their weight in kilograms.
Height | Once every two weeks for 105 days
  The participants were measured for their height in cm.
Body Mass Index (BMI) | Once every two weeks for 105 days
  The measurement of weight and height were combined into BMI and expressed in kg/m^2
Arm circumference | Once every two weeks for 105 days
  The participants were measured for their arm circumference in cm.
Head circumference | Once every two weeks for 105 days
  The participants were measured for their head circumference in cm.
Subcutaneous fat thickness | Once every two weeks for 105 days
  The participants were measured for their subcutaneous fat thickness in mm.
Triceps thickness | Once every two weeks for 105 days
  The participants were measured for their triceps thickness in mm.
Medical check up | Once every two weeks for 105 days
  An on-site medical professional will check the health condition of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Endang Sutriswati Rahayu, Prof. Dr. Ir, Principal Investigator — Gadjah Mada University
Locations (10):
- Indonesia (10):
  - PAUD Hiber Rotowijayan, Yogyakarta, Special Region of Yogyakarta
  - Paud Kunir Ceria Tegalgendu Kotagede, Yogyakarta, Special Region of Yogyakarta
  - Puskesmas Mlati 2, Yogyakarta
  - Paud Bodeh, Yogyakarta
  - Paud Gamping Lor, Yogyakarta
  - Paud Matahari Mejing 3, Yogyakarta
  - Paud Pereng Dawe, Yogyakarta
  - Paud Pereng Kembang, Yogyakarta
  - Paud Sembung, Yogyakarta
  - Paud Sumber, Yogyakarta

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers. During the screening period, all participants' guardian signed informed consent that states the data will not be shared to others aside from the current researcher and sponsors in the study.